CLINICAL TRIAL: NCT04651803
Title: Factors Associated With Unfavorable Outcome in Traumatic Brain Injury Elderly Patients. A Retrospective Multicenter Study
Brief Title: Outcome in Traumatic Brain Injury Elderly Patients
Status: Completed | Type: Observational
Sponsor: Association pour la Recherche en Aanesthésie Réanimation Digestive (Other)
Responsible Party: Principal Investigator, SEGUIN Philippe, President, Association pour la Recherche en Aanesthésie Réanimation Digestive
Other Study IDs: ATLANREA
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Traumatic brain injury patients: Traumatic brain injury patients admitted in intensive care unit.

SUMMARY:
In patients suffering from traumatic brain injury (TBI), the study's purpose was to determinate factors associated with mortality and poor functional outcome at 3 months in patients aged ≥ 65 hospitalized in ICU and to compare outcome at 3 months between younger patients (18-64 years) vs older patients (≥65 years).

Traumatic brain injury is a common cause of hospitalization for trauma and accounting for roughly 37% of all injury-related death in Europe. This was particularly true for patients ≥ 65 years old and in the most severe case(Glasgow coma score ≤ 8) with mortality rates between 31 to 51%. Over time, epidemiological patterns of TBI are changing. Indeed, in high-income countries, overall incidence is steadily decreasing, but increasing in elderly population with falls becoming the leading cause of TBI. In parallel, the World Population Ageing 2019 report of the Population Division of the United Nations Department of Economic and Social Affairs reported 703 (9%) million persons aged ≥65 years in the global population and that this proportion is projected to rise further to 16 % in 2050. Accordingly, we could expect that TBI in elderly would be increasing and could explain why mortality did not improved in the latest decades.

In a study performed in three neuro-intensive care unit (ICUs) from 1997 to 2007, 6-month mortality in patients aged of 70-79 and ≥ 80 years was 59% and 79%, respectively. In severe elderly (≥ 65 years) TBI patients admitted in ICU, hospital and 6-month mortality was 64.6% and 72.9%, respectively. Beyond mortality, TBI can lead to poor functional neurologic outcome and elderly patients are more prone to survive with disabilities according to a higher rate of comorbidities, frequent use of oral anticoagulants and/or antiplatelet and/or previous brain disorders. In patients hospitalized in ICU, age (> 59 years) was the strongest parameter associated with an unfavorable outcome including death, vegetative state and severe disability, at 6 month. Moreover, TBI elderly patients (≥ 65 years) had worse functional outcome at discharge than younger patients. Identifying elderly patients who may benefit from ICU remained challenging, since there is no consensual guideline of triage. Traumatic brain-injured patients are particularly concerned by this issue. Nevertheless, few data are available related to outcome in elderly TBI patients requiring ICU.

DETAILED DESCRIPTION:
The investigators conducted a multicentre, retrospective, observational study from April 2013 to February 2019 in the surgical ICUs of 5 level 1 Trauma centers in France. The investigators collected data from the "regional intensive care network of the great west of france" (AtlanRéa) database. The AtlanRéa database registers prospectively and consecutively numerous informations about brain injury and trauma patients hospitalized in ICUs, in order to provide epidemiologic informations for this population. Data were collected by clinical research assistants in each participating ICU, using an electronic case report form. The investigators assessed data regarding outcomes after discharge from ICUs through phone interview led by dedicated clinical research assistants.

The following data were entered in the database: Age, gender and body mass index, previous medical history, and more specifically the presence of cardiac insufficiency, chronic renal failure defined as an estimated glomerular filtration rate less than 60 ml/min.1.73 m-1, chronic respiratory illness, neurologic background, diabetes, neoplasia history, previous TBI, active smoking and chronic alcoholism. Mechanism of injury (domestic accident, road traffic crash, fall from heights or others). The Glasgow Coma Score (GCS) score determinates in the prehospital setting or at admission at hospital before intubation and/or sedation, and the presence of at least one nonreactive and dilated pupil at the initial management. Severity of illness according to the Simplified Acute Physiology Score II (SAPS II) the Sequential Organ Failure Assessment (SOFA) score, and the Injury Severity Score (ISS). The investigators also specified the severity of TBI by the abbreviated Injury Score (AIS) and reported the associated injuries from 5 territories (face, chest, abdomen, extremity (including pelvis) and external). Initial CT-scan was classified according to the Marshall classification in six categories (Diffuse injury I, II, III, IV, evacuated mass (V) and non-evacuated mass lesion (VI)).

The following data during the patients' hospitalization are also entered in the database: use of an intracranial pressure (ICP) catheter, occurrence of intracranial hypertension (defined as an ICP above 20 mmHg in absence of confounding factors), and use of barbiturates and/or osmotherapy, decompressive craniectomy, and other neurosurgical procedure. The occurrence of intercurrent events occurring during ICU stay, including infections, Acute Respiratory Distress Syndrome (ARDS), need of vasopressor drugs, acute renal failure, thrombophlebitis, pulmonary embolism, hemorrhage, infection and tracheostomy. The investigators specified the need for intubation and durations of mechanical ventilation, central venous catheterism and vasopressor. The investigators also recorded the decision in ICU to withdraw or withhold life support.

The length of stay in ICU, ICU and 3-month mortalities and patient outcome were assessed using the Glasgow Outcome Scale Extended (GOSE) score at 3 months. The investigators dichotomized the GOSE score between the four lower values (corresponding to unfavorable outcome- GOSE 1 to 4) and the four upper values (corresponding to favorable outcome- GOSE 5 to 8).

Statistical Analysis All statistical analysis will be performed using R software 3.3.1 (package pROC) and SAS 9.1 Statistical Software (SAS Institute, Cary, NC, USA). For quantitative continuous variables, position and dispersion parameters (mean, standard deviation, median, interquartile range) will be calculated. For qualitative variables, proportion rates will be calculated. For groups' comparison, we used independent-samples t-tests for normally distributed continuous variables, and Mann-Whitney U-tests for non-normally distributed continuous variables. Χ² tests will be performed for categorical variables. To build the model for multivariate analysis, the investigators selected among the variables with a p ≤ 0.20 according to the univariate analysis. The investigators performed logistic regression model to identify factors associated with in-ICU mortality and dichotomized GOSE score at 3 months. The Odds Ratios (ORs) and 95% confidence intervals (CI) will be calculated. For continuous variables, diagnosis of log linear behavior was established, and if not confirmed, the variable will be divided into categories and treated as categorical variables. Model's fit will be assessed by checking residual plots and Cook's distance. The calibration of the model will be tested by Goodness of Fit Hosmer-Lemeshow test. A p ≤0.05 will be considered statistically significant for all the comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury
* Aged at least 18 years,
* Hospitalized in intensive care unit

Exclusion Criteria:

* Patients who die within 24h of hospitalization
* Patients initially resuscitated awaiting for organ donation
* Refusal for study participation expressed by the patient or relatives.
* Missing data related to the main objective of the study (outcome at 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 1633 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Outcome was assessed using the Glasgow Outcome Scale Extended (GOSE) score | GOSE score at 3 months.
  We dichotomized the GOSE score between the four lower values (corresponding to unfavorable outcome- GOSE 1 to 4) and the four upper values (corresponding to favorable outcome- GOSE 5 to 8).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Seguin, MD, PhD, Principal Investigator — AtlanRéa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roozenbeek B, Maas AI, Menon DK. Changing patterns in the epidemiology of traumatic brain injury. Nat Rev Neurol. 2013 Apr;9(4):231-6. doi: 10.1038/nrneurol.2013.22. Epub 2013 Feb 26. PMID 23443846
- [Background] Stocchetti N, Paterno R, Citerio G, Beretta L, Colombo A. Traumatic brain injury in an aging population. J Neurotrauma. 2012 Apr 10;29(6):1119-25. doi: 10.1089/neu.2011.1995. Epub 2012 Apr 2. PMID 22220762
- [Background] Maiden MJ, Cameron PA, Rosenfeld JV, Cooper DJ, McLellan S, Gabbe BJ. Long-Term Outcomes after Severe Traumatic Brain Injury in Older Adults. A Registry-based Cohort Study. Am J Respir Crit Care Med. 2020 Jan 15;201(2):167-177. doi: 10.1164/rccm.201903-0673OC. PMID 31657946
- [Background] Gardner RC, Dams-O'Connor K, Morrissey MR, Manley GT. Geriatric Traumatic Brain Injury: Epidemiology, Outcomes, Knowledge Gaps, and Future Directions. J Neurotrauma. 2018 Apr 1;35(7):889-906. doi: 10.1089/neu.2017.5371. Epub 2018 Feb 15. PMID 29212411
- [Background] Lim XT, Ang E, Lee ZX, Hajibandeh S, Hajibandeh S. Prognostic significance of preinjury anticoagulation in patients with traumatic brain injury: A systematic review and meta-analysis. J Trauma Acute Care Surg. 2021 Jan 1;90(1):191-201. doi: 10.1097/TA.0000000000002976. PMID 33048909
- [Background] Susman M, DiRusso SM, Sullivan T, Risucci D, Nealon P, Cuff S, Haider A, Benzil D. Traumatic brain injury in the elderly: increased mortality and worse functional outcome at discharge despite lower injury severity. J Trauma. 2002 Aug;53(2):219-23; discussion 223-4. doi: 10.1097/00005373-200208000-00004. PMID 12169925
- [Background] De Bonis P, Pompucci A, Mangiola A, Paternoster G, Festa R, Nucci CG, Maviglia R, Antonelli M, Anile C. Decompressive craniectomy for elderly patients with traumatic brain injury: it's probably not worth the while. J Neurotrauma. 2011 Oct;28(10):2043-8. doi: 10.1089/neu.2011.1889. Epub 2011 Aug 29. PMID 21639728
- [Background] Pettigrew LE, Wilson JT, Teasdale GM. Reliability of ratings on the Glasgow Outcome Scales from in-person and telephone structured interviews. J Head Trauma Rehabil. 2003 May-Jun;18(3):252-8. doi: 10.1097/00001199-200305000-00003. PMID 12802167
- [Result] Majdan M, Plancikova D, Brazinova A, Rusnak M, Nieboer D, Feigin V, Maas A. Epidemiology of traumatic brain injuries in Europe: a cross-sectional analysis. Lancet Public Health. 2016 Dec;1(2):e76-e83. doi: 10.1016/S2468-2667(16)30017-2. Epub 2016 Nov 29. PMID 29253420
- [Derived] Launey Y, Coquet A, Lasocki S, Dahyot-Fizelier C, Huet O, Le Pabic E, Roquilly A, Seguin P. Factors associated with an unfavourable outcome in elderly intensive care traumatic brain injury patients. a retrospective multicentre study. BMC Geriatr. 2022 Dec 30;22(1):1004. doi: 10.1186/s12877-022-03651-x. PMID 36585608
- See also: World Population Ageing 2019 — http://www.un.org/en/development/desa/population/publications/pdf/ageing/WorldPopulationAgeing2019-Highlights.pdf